CLINICAL TRIAL: NCT02474420
Title: The Use of the Calcium Channel Blocker Amlodipine as an Adjuvant Treatment to Iron Chelation for the Prevention of Iron Overload Cardiomyopathy in Patients With Thalassemia
Brief Title: Amlodipine as Adjuvant Treatment to Iron Chelation for Prevention of Cardiac Iron Overload in Thalassemia Patients
Acronym: CANALI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kevin H.M. Kuo, MD, MSc, FRCPC (Other)
Responsible Party: Sponsor-Investigator, Kevin H.M. Kuo, MD, MSc, FRCPC, Assistant Professor, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CANALI
Record Dates: First submitted 2015-06-11; First posted 2015-06-17 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Beta-Thalassemia; Iron Overload
MeSH Terms: conditions — beta-Thalassemia; Iron Overload | interventions — Amlodipine; Deferasirox

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deferasirox (Active Comparator): deferasirox iron chelation therapy and standard of care by the treating physician
  Interventions: Drug: Deferasirox
- Deferasirox plus amlodipine (Experimental): deferasirox iron chelation therapy with amlodipine
  Interventions: Drug: Amlodipine; Drug: Deferasirox

INTERVENTIONS:
Drug: Amlodipine — amlodipine titrated up to 10 mg daily or maximum tolerated dose, whichever comes first
  Arms: Deferasirox plus amlodipine
Drug: Deferasirox — Deferasirox administered per standard of care by the treating physician

SUMMARY:
This is a randomized, open label, two arms superiority trial of a representative population of patients with a primary diagnosis of transfusion dependent thalassemia with evidence of moderate cardiac iron overload, defined as an average T2* MRI parameter at the mid inter-ventricular septum between 10 and 20ms.

DETAILED DESCRIPTION:
Selection of Study Population: The study will enroll 60 adult subjects with transfusion dependent thalassemia receiving deferasirox iron chelation therapy. All eligible subjects will be asked to provide informed consent before participating in the study.

Randomization: Subjects will be randomized in a 1:1 ratio to either continuation of their DFX (control arm) or a combination of DFX plus amlodipine (amlodipine arm).

Treatment: Subjects randomized to the amlodipine arm will receive open label medication (amlodipine) starting at 2.5mg/day and up-titrated by 2.5mg every 7-14 days with the goal of reaching 10mg/day. DFX dose in either arm will not be adjusted unless it was deemed unsafe to remain on the same dose of DFX by the treating physician (significant side effects, lack of efficacy or over-chelation) or T2* drops below 8 ms.

Safety Assessment: Weekly or fortnightly amlodipine titration will be conducted by the research physician in-clinic, based on blood pressure, tolerability, and presence or absence of side-effects.

Adverse Events will be assessed at every visit after the first dose through to the last subject visit.

Efficacy Assessment: the efficacy of amlodipine combined to standard chelation therapy will be assessed by cardiac T2*MRI, done at baseline and 12 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of transfusion-dependent Thalassemia being followed by a thalassemia comprehensive care clinic Age 18 or older
* Taking deferasirox and on a stable dose for >3 months
* Evidence on cardiac MRI of mild to moderate cardiac iron overload (T2*<20ms but ≥10ms) as measured within 3 months prior to randomization. If a recent cardiac MRI has not been obtained, patients who otherwise meet all eligibility criteria and provide appropriate consent will undergo a cardiac MRI to confirm eligibility
* Preserved left ventricular ejection fraction (LVEF) >55% as measured by cardiac MRI. If a recent cardiac MRI has not been obtained, patients who otherwise meet all eligibility criteria and provide appropriate consent will undergo a cardiac MRI to confirm eligibility.
* Agreeable to use an approved method of contraception if female of childbearing potential for the entire duration of the study.

Exclusion Criteria:

* Serum ferritin < 500 ng/mL at screening
* Liver iron concentration > 30 mg/g dw as measured by liver R2 MRI (FerriScan)
* Congestive heart failure
* Severe refractory Hypotension (less than 90 mmHg systolic)
* Currently taking any calcium channel blockers
* Pregnancy or nursing (a negative HCG (pregnancy) test must be obtained prior to randomization)
* As a result of medical review, physical examination or screening investigations, the Principal Investigator (PI) considers the subject unfit for the study
* No fixed address
* Hypersensitivity to amlodipine or other dihydropyridines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac T2* | 12 months following randomization
  Change in cardiac T2* as determined by MRI

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction | 12 months following randomization
  Change in left ventricular ejection fraction (in %) as determined by MRI
Number of Participants with Adverse Events | 12 months following randomization

CONTACTS AND LOCATIONS:
Overall Officials: Kevin HM Kuo, MD MSc FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597